CLINICAL TRIAL: NCT06519565
Title: Clinical Study on the Safety and Efficacy of PRG-1801 for the Treatment of Recurrent/Refractory Primary Immune Thrombocytopenia (ITP)
Brief Title: Safety and Efficacy of PRG-1801 in Recurrent/Refractory Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Shenzhen Pregene Biopharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG1801E13
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-12

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: PRG-1801 Injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRG-1801(BCMA-targeting CAR-T Cells) (Experimental): The study was structured into two distinct phases: the dose exploration phase and the dose expansion phase. During the dose exploration phase, three dosage levels were established-100x10^6 CAR-T and 200x10^6 CAR-T-with each dosage group comprising 3 to 6 subjects with Immune Thrombocytopenia (ITP). If dose-limiting toxicity (DLT) was observed in one out of three subjects within any dosage group, an additional three subjects were enrolled at the same dosage level. Should DLT be present in two or more out of six subjects, considerations for dose reduction or potential study discontinuation were made.
  Upon determining the safe and effective fixed dose of PRG-1801 during the dose exploration phase, the study progressed to the dose expansion phase. This subsequent phase involved enrolling an additional 3 to 6 subjects at the established fixed dose. The aim was to further assess and confirm the safety and efficacy of this specific dose for treating ITP.
  Interventions: Drug: PRG-1801

INTERVENTIONS:
Drug: PRG-1801 — PRG-1801 is a chimeric antigen receptor T-cell (CAR-T) therapy targeting BCMA. Participants will undergo leukapheresis to collect mononuclear cells for PRG-1801 manufacturing. Prior to infusion, patients receive lymphodepletion with cyclophosphamide (250-300 mg/m2/day) and fludarabine (25-30 mg/m2/day) for 3 days. PRG-1801 is then administered as a single intravenous infusion at one of three dose levels: 100×10^6, or 200×10^6 CAR-T cells. Premedication with antipyretics and antihistamines is given 30-60 minutes before infusion. The infusion rate is 2-5 ml/min. Patients are monitored for safety and efficacy for up to 24 months post-infusion. Some patients may be eligible for a second infusion if they respond initially but later relapse.
  Other Names: BCMA-targeting CAR-T Cells

SUMMARY:
This is a single center, open-label, 3+3 dose escalation, early phase 1 study to evaluate the safety, tolerability, and preliminary efficacy of PRG-1801 for patients with relapsed/refractory immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This investigator-initiated clinical study aims to evaluate PRG-1801, a BCMA-targeted CAR-T cell therapy, in patients with relapsed refractory immune thrombocytopenia (ITP). The study employs a dose-escalation design to assess safety, tolerability, and preliminary efficacy.

Approximately 1 sites are planned to be selected for the clinical trial. The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 100×10^6, and 200×10^6 CAR-T cells groups in order of sequence. And the subjects will undergo leukapheresis, lymphodepletion pre-treatment, and a single infusion of PRG-1801. Dose escalation will follow 3 + 3 design and 3-6 subjects in each group will complete a single dose. Within the same dose group, the next subject will be administered after the previous subject has completed at least 14 days of safety observation. After the last subject in each dose group has completed the dose-limiting toxicity (DLT) assessment window of 28 days after single dose, the enrollment and treatment for the next dose group may be initiated after the Safety Review Committee (SRC) agrees to enter the next dose group based on clinical safety data assessment.

When DLT occurs in 1 of 3 subjects in a dose group, 3 additional subjects in the same dose group will be required (up to 6 subjects in the dose group have completed DLT assessment): if no DLT occurs in the additional 3 subjects, dose escalation will continue; if 1 of the 3 additional subjects experiences one DLT, dose escalation will be discontinued; if more than 1 of the 3 additional subjects experiences DLTs, dose escalation will be discontinued, and 3 additional subjects will be required to be enrolled at one lower dose level for DLT assessment. After the end of escalation for the maximum dose group, if no MTD is observed, the highest dose level is defined as the MTD

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years, regardless of gender.
* 2. Clinically diagnosed with primary immune thrombocytopenia for at least 6 months, with a platelet count <30×10^9/L within 48 hours before participating in the study.
* 3. Positive for anti-platelet glycoprotein autoantibodies (such as GPIIb/IIIa).
* 4. Previously received first-line and/or second-line ITP treatment (first-line treatment includes: corticosteroids or immunoglobulins; second-line treatment includes thrombopoietin receptor agonists (such as eltrombopag, romiplostim) and/or rituximab, etc.), but the treatment was ineffective (platelet count <30×10^9/L after treatment, or platelet count did not increase to twice the baseline value, or there was bleeding), or relapsed after effective treatment (platelet count dropped below 30×10^9/L after effective treatment, or dropped to less than twice the baseline value, or bleeding symptoms occurred) or difficult to maintain after stopping TPO receptor agonists.
* 5. Basic normal function of important organs:

  * Echocardiography indicates an ejection fraction ≥50%, and the electrocardiogram shows no significant abnormalities.
  * Creatinine clearance rate (CrCl) (Cockcroft-Gault formula) ≥30 mL/min.
  * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤3.0× the upper limit of normal (ULN).
  * Total bilirubin (TBIL) and alkaline phosphatase (AKP or ALP) ≤2.0×ULN (Gilbert's syndrome ≤ 3.0×ULN).
  * Absolute lymphocyte count (ALC) ≥0.5×10^9/L; absolute neutrophil count (ANC) ≥1×10^9/L; hemoglobin (Hb) ≥60 g/L; platelet count ≥10×10^9/L.
  * Blood oxygen saturation >92%.
* 6. Meet the standards for apheresis or venous blood collection, and have no contraindications to cell collection.
* 7. Men of reproductive potential and women of childbearing age must agree to use effective contraception from the signing of the informed consent form until 1 year after the use of the study drug. Blood pregnancy tests for women of childbearing age must be negative at screening and before cell infusion, and they must not be breastfeeding.
* 8. The participant or their guardian agrees to participate in this clinical trial and signs the informed consent form (ICF), indicating their understanding of the purpose and procedures of this clinical trial and their willingness to participate in the study.

Exclusion Criteria:

* 1. Thrombocytopenia caused by myelodysplastic syndromes, early aplastic anemia, atypical aplastic anemia, thrombotic thrombocytopenic purpura, etc.
* 2. Bone marrow examination during the screening period suggests myelofibrosis MF≥2 (European consensus scoring standard Thieleja2005) or bone marrow examination indicates the presence of primary diseases other than ITP that can cause thrombocytopenia.
* 3. Allergic history to any component in the cell product.
* 4. Suffering from any of the following heart diseases:

  * Congestive heart failure of NYHA class III or IV.
  * Myocardial infarction or coronary artery bypass grafting (CABG) or coronary stent implantation within ≤6 months before signing the ICF.
  * Clinically significant ventricular arrhythmias, or history of unexplained syncope (excluding vasovagal syncope or dehydration).
  * Severe non-ischemic cardiomyopathy history.
* 5. Malignant tumors within the past 3 years before screening, except for the following: malignant tumors that have been treated radically and have no known active disease for ≥3 years before enrollment; or well-treated non-melanoma skin cancer with no evidence of disease.
* 6. Symptomatic deep vein thrombosis or pulmonary embolism within the past 6 months or currently requiring anticoagulant therapy.
* 7. Participation in other interventional clinical studies within 1 month before screening.
* 8. Vaccination with attenuated live vaccines within 4 weeks before screening.
* 9. Stroke or epileptic seizure within 6 months before signing the ICF (excluding old lacunar cerebral infarction).
* 10. The following treatments before CAR-T reinfusion: immunosuppressive treatment within 3 days; use of prednisone (or equivalent drugs) at a dose >10mg/day within 3 days.
* 11. The following treatments before CAR-T reinfusion: treatment with B-cell depleting agents such as rituximab within 24 weeks (unless B cells have recovered); immunoglobulin reinfusion treatment within 4 weeks.
* 12. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer detection exceeds the normal range; positive for hepatitis C virus (HCV) antibody and peripheral blood hepatitis C virus (HCV) RNA titer detection exceeds the normal range; positive for human immunodeficiency virus (HIV) antibody; positive syphilis test.
* 13. Other conditions deemed unsuitable for participation in the study by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | Up to 28 days post-infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The safe dosage for a single infusion of PRG-1801 | Up to 28 days post-infusion
  The safe PRG-1801 infusion dosage for ITP patients will be evaluated by comprehensively assessing the complete response (CR) rate and the incidence of adverse events (AEs).

SECONDARY OUTCOMES:
Complete response (CR) rate or Response (R) rate of administering PRG-1801 in the treatment of relapsed/refractory ITP | At Day 28, Month 2, Month 3, Month 6,Month 9, Month 12, Month 18, and Month 24 post-infusion
  CR is defined as platelet count ≥100×10^9/L. R is defined as platelet count ≥30×10^9/L and at least doubling from baseline, without active bleeding.
The proliferation rate and persistence time of CAR-T cells | At baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24 post-infusion
  Evaluation of CAR-T cell expansion and persistence through measurement of CAR copy number in peripheral blood
Concentration of serum sBCMA, immunoglobulins (IgG, IgM, IgA), and anti-platelet glycoprotein autoantibodies | At baseline, Day 28, Month 2, Month 3, Month 6,Month 9, Month 12, Month 18, and Month 24 post-infusion
  Pharmacodynamics of PRG-1801 were assessed by evaluating changes from baseline in serum sBCMA, immunoglobulins (IgG, IgM, IgA), and anti-platelet glycoprotein autoantibodies

OTHER OUTCOMES:
Evaluation of incidence of Treatment-related Adverse Events and Complete response rate or Response rate of repeated PRG-1801 infusion | Up to 24 months after second infusion
  The evaluation metrics are the same as those for the primary and secondary outcome measures of single infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Ph.D&M.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No